CLINICAL TRIAL: NCT06066073
Title: Pain Perception and Emotional Changes On The Relationships Between Dental Anxiety And Olfaction: A Double-blinded Randomized Control Trial
Brief Title: "Pain and Emotional Changes on Relationships Between Anxiety and Olfaction"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Qassim University (Other)
Responsible Party: Principal Investigator, Ghada Amin Khalifa, PhD, Professor of Maxillofacial Surgery and Diagnostic Science, Qassim University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: EA/3006/2018
Record Dates: First submitted 2021-05-18; First posted 2023-10-04 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-09

CONDITIONS: Anxiety
Keywords: Pain; Anxiety; Fear; Stress
MeSH Terms: conditions — Anxiety Disorders; Pain | interventions — lavender oil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lavender group (Experimental): Patients who were included in this group were subjected to vapors of the lavender oil in waiting rooms, during dental therapy, and on day after dental procedures
  Interventions: Drug: Lavender Oil
- Control group (Placebo Comparator): Patients who were included in this group were subjected to vapors of distal water in waiting rooms and during dental therapy
  Interventions: Drug: Distal Water

INTERVENTIONS:
Drug: Lavender Oil — Twenty drops of lavender oil was added the distal water which fill the vaporizer which were placed in the waiting room. The patients inhaled the vapors of the lavender oil 20 minutes before starting the dental procedures
  Other Names: Lavandula angustifolia.
  Arms: Lavender group
Drug: Distal Water — The patients inhaled vapors of the distal water in the waiting room 20 minutes before starting dental procedures
  Other Names: Deionized water
  Arms: Control group

SUMMARY:
Introduction: This prospective study aimed to assess the impact of olfaction on providing positive emotional responses and reducing dental anxiety and pain.

Material: A randomized double-blinded controlled study was enrolled on female patients. The olfaction was stimulated via lavender essential oils. Patients were divided into lavender and control groups. Patients in lavender group inhaled 2 % lavender vapors. In control group, patients inhaled distal water vapors. The variables included pain, anxiety, and vital signs. Anxiety was measured through Modified Dental Anxiety Scale (MDAS) and Speilberger State-Trait Anxiety Inventory (STAI) questionnaires. Pain was evaluated through visual analog scales (VAS). Vital signs included the systolic (SBP) and diastolic blood pressure (DBP), heart rate (HR), respiratory rate (RR), and oxygen saturation (Spo2). All variables were assessed before the intervention, 20 minutes after inhalation of vapors, and at the end of dental settings. The last evaluation was on the day after visits. P-values < 0.05 were considered significant.

DETAILED DESCRIPTION:
ABSTRACT:

Background: The purpose of the study was to determine to what extent olfactory aromatherapy reduces the intensity of dental pain and the level of dental anxiety. It also attempted to corelate between olfactory aromatherapy, stages of dental visits, and various dental procedures.

Methods: Female patients were enrolled in a randomized controlled study. Olfactory aromatherapy was performed using lavender oils. Patients were randomly assigned to one of two groups: the lavender group, in which patients inhaled 2% lavender vapors, and the control group, in which patients inhaled water vapors. Pain score, anxiety score, and changes in vital signs were among the predictable variables. Anxiety and pain were assessed using the Modified Dental Anxiety Scale (MDAS), Speilberger State-Trait Anxiety Inventory (STAI), and visual analog scales (VAS). The vital signs were systolic (SBP) and diastolic (DBP), heart rate (HR), respiratory rate (RR), and oxygen saturation (Spo2). Variables were evaluated before inhalations, 20 minutes after inhalations, at the end of settings, and on the following day.

ELIGIBILITY:
Inclusion Criteria:

* Adult females over 18 years,
* Attending morning sessions of clinics (9 am),
* Liable for administration of local anesthesia, tooth preparation either for:

  1. Filling procedures or crown preparations
  2. Endodontic treatment
  3. Teeth extraction
  4. Eubgingival scaling

Exclusion Criteria:

* Males
* Females who had:

  1. Allergies
  2. Bronchial asthma
  3. Common cold
  4. Pulmonary diseases
  5. Migraine
* Females who taking:

  1. Antidepressants
  2. Anxiolytic drugs
  3. Opioids
  4. Other medications that affect emotional responses
* Pregnant females

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 350 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
Anxiety score | 20 minutes after exposure
  Measured by Dental anxiety was measured by the Modified Dental Anxiety Scale (MDAS) questionnaire
Pain Score | 20 minutes after exposure
  Measured by a visual analog scale (VAS).These pain scales give people a simple way to rate their pain intensity using a verbal or visual descriptor of their pain. Some examples would be the words "mild," "discomforting," "distressing," "horrible," and "excruciating."

SECONDARY OUTCOMES:
Blood pressure | 20 minutes after exposure
  The patients were asked to stand up straight, and the sphygmomanometer cuff was inserted around their upper left arms, with a 2.5-inch distance between the antecubital fossa of the arm and the lower edge of the cuff. The blood pressure was measured after the stethoscope was placed over the brachial artery

CONTACTS AND LOCATIONS:
Overall Officials: Ghada A Khalifa, Professor, Study Director — College of Dentistry, Qassim University, Saudi Arabia
Locations (1):
- College of Dentistry, Qassim University, Buraidah, Al-Qassim Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No